CLINICAL TRIAL: NCT04297488
Title: Effect and Safety of Probiotic Supplementation in Immune Non-responders With HIV-1 Infection
Brief Title: Probiotic Supplementation for Those Immune Non-responders With HIV-1 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CACTGUT20
Record Dates: First submitted 2018-06-08; First posted 2020-03-05 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: HIV-infection/Aids
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INR(oral probiotic capsules containing 3 billion Bifidobacterium and 1 billion Lactobacillus) (Experimental): Participants will receive oral probiotic capsules containing 3 billion Bifidobacterium and 1 billion Lactobacillus once daily for 6 months.
  Interventions: Dietary Supplement: Bifidobacteria and Lactobacilli triple viable capsules

INTERVENTIONS:
Dietary Supplement: Bifidobacteria and Lactobacilli triple viable capsules — Bifidobacteria and Lactobacilli triple viable capsules (provided by Shenzhen Wan he Pharmaceutical Co., Ltd., China) are bilayer mini pellets and are resistant to gastric acid. So Bifidobacterium billion Lactobacillus can only be released in intestine. Participants will take 1.27g (contain 3 billion Bifidobacterium and 1 billion Lactobacillus) once daily.

SUMMARY:
Gut bacterial community diversity and composition, immune recovery and activation in peripheral plasma/mucosa, plasma levels of gut damage, microbial translocation and inflammation at baseline and after 6 months of receiving intervention will be analyzed.

DETAILED DESCRIPTION:
Up to 25% of HIV-infected individuals receiving antiretroviral treatment demonstrate suboptimal blood cluster of differentiation 4（CD4） recovery despite effective viral suppression; this "immunologic non-responder" (INR) phenotype is associated with increased immune activation and with higher rates of AIDS and non-AIDS related conditions, and death. Poor gut integrity, increased microbial translocation, and reduced CD4 T-cell trafficking to the gut could be a source of ongoing inflammation in INR individuals. Researches have shown that the gut microbiota compositions are different in INRs and immunological responders (IRs). Probiotics, by modulation of gut microbiota, can help induce epithelial healing and prevent bacterial translocation. Probiotic supplementation, therefore, may be a nutritional target for INRs by boosting CD4 cell counts. We design a prospective, case-control, self-contrast study to explore the efficacy and safety of probiotic supplementation in INRs. Participants will receive oral probiotic containing 3 billion Bifidobacterium and 1 billion Lactobacillus once daily. Gut bacterial community diversity and composition, immune recovery and activation in peripheral plasma/mucosa, plasma levels of gut damage, microbial translocation and inflammation at baseline and after 6 months of receiving intervention will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* 18-65 years old
* On antiretroviral therapy (>2 years)
* Ability to provide informed consent
* Undetectable plasma HIV-1 viral load for the past 2 years
* CD4 T-cell count <350/mm3 for the last 2 years
* No history of gastrointestinal diseases

Exclusion Criteria:

* Administration of antibiotics, probiotics, or prebiotics or experience of diarrhea within the previous 3 months;
* Administration of anti-inflammatory drugs, corticosteroids, immunosuppressive drugs, immunomodulator within the previous 3 months;
* Severe organ dysfunction
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Immune recovery and activation | Changes from baseline to 6 months
  CD4+ T-cell and cluster of differentiation 8（CD8）+ T-cell counts, CD4/CD8 ratio, cluster of differentiation 38（CD38）+/ human leukocyte antigen(HLA）-HLA class II(DR)+ CD8+/CD4+ T cell ratio

SECONDARY OUTCOMES:
Plasma levels of gut damage, microbial translocation and inflammation | Changes from baseline to 6 months
  interleukin(IL)-8, IL-1β, IL-6, tumor necrosis factor(TNF)-α, C reactive protein(CRP), D-dimer, Intestinal fatty aid binding protein(I-FABP), lipopolysaccharide(LPS) , lipopolysaccharide-binding protein(LBP), sCD14, sCD40L, and Kynurenine/Tryptophan ratio
Blood viral load | Changes from baseline to 6 months
  HIV-RNA
Metabolic measurements from blood plasma | Changes from baseline to 6 months
  Vitamin D, glucose and insulin, and lipid profiling
Feasibility, safety, tolerability, adherence, and acceptability of study product and procedures | Changes from baseline to 6 months
  Based on patients' description and intervention-related adverse events
Gut bacterial community diversity and composition | Changes from baseline to 6 months
  Bacterial community diversity and composition determined by 16S ribosomal ribonucleic acid(rRNA) gene sequencing of fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: WEI Lyu, Principal Investigator — Department of Infectious Diseases, PekingUMCH
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No